CLINICAL TRIAL: NCT07354984
Title: A Single-Arm Phase II Clinical Study of Docetaxel Combined With Nimotuzumab and Pucotenlimab as Second-Line and Beyond Therapy for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Acronym: PIONEER-HN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Biotech Pharmaceutical Co., Ltd. (Other); Lepu Biopharma Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chen Chunyan, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-390
Record Dates: First submitted 2025-12-31; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: R/M HNSCC; Second-line therapy; Immune Checkpoint Inhibitors; Salvage Therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy, Combination; Docetaxel; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): This single-arm phase II study evaluates the efficacy and safety of docetaxel, nimotuzumab, and pucotenlimab combination therapy as second- or later-line treatment in patients with recurrent or metastatic head and neck squamous cell carcinoma (R/M HNSCC) who have failed prior PD-1/PD-L1 inhibitors and platinum-based chemotherapy. All enrolled patients must have unresectable, radiotherapy-ineligible R/M HNSCC, and ≤2 prior lines of therapy. Following screening and informed consent, treatment endpoints are defined from first dose until disease progression, death, intolerable toxicity, consent withdrawal, new anti-tumor therapy initiation, or other protocol-specified discontinuation criteria.
  Interventions: Drug: Drug Combination Therapy

INTERVENTIONS:
Drug: Drug Combination Therapy — [Docetaxel 75mg/m2 + Nimotuzumab 400mg + Pucotenlimab 200mg], intravenous infusion, Day 1, every 3 weeks, for 4-6 cycles (exact number determined by investigator assessment).
  Maintenance Regimen: [Nimotuzumab 400mg + Pucotenlimab 200mg], intravenous infusion, Day 1, every 3 weeks, until protocol-defined treatment endpoints are reached.
  Maintenance Therapy Eligibility: Subjects who meet both criteria after the last induction cycle: No disease progression confirmed by imaging and investigator assessment, and/or absence of intolerable toxicity.
  Other Names: Docetaxel; Nimotuzumab; Pucotenlimab

SUMMARY:
This study is a single-arm Phase II trial designed to evaluate the efficacy and safety of Docetaxel, Nimotuzumab, and Pucotenlimab combination therapy in patients with recurrent or metastatic head and neck squamous cell carcinoma who have failed prior PD-1/PD-L1 inhibitor and platinum-based therapies, for second-line and later-line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1, with no deterioration within 2 weeks prior to enrollment.
2. Age ≥ 18 years and ≤ 75 years
3. Patients with pathologically and/or radiologically confirmed recurrent or metastatic head and neck squamous cell carcinoma (including oral cavity, oropharynx, hypopharynx and larynx), who have previously failed treatment with PD-1 (L1) inhibitors and platinum-based drugs. The two types of drugs could be administered as a first-line combination regimen or sequential therapy, with the number of prior treatment lines not exceeding two. If disease progression occurs during neoadjuvant therapy, concurrent chemoradiotherapy or adjuvant therapy, or within 6 months after the discontinuation of such treatment, the medications used during neoadjuvant therapy, concurrent chemoradiotherapy or adjuvant therapy (including platinum-based drugs, anti-EGFR monoclonal antibodies, PD-1 (L1) inhibitors, etc.) shall be regarded as first-line treatment. Discontinuation or dose reduction of one drug during treatment, or replacement of platinum-based drugs, fluorouracil-based drugs or PD-1 (L1) inhibitors without disease progression shall be counted as the same line of treatment.
4. At least one radiologically measurable lesion according to RECIST v1.1
5. Assessed by the investigator as not amenable to local therapy (e.g., surgery ± radiotherapy)
6. PD-L1 Combined Positive Score (CPS) ≥ 1
7. Adequate organ function
8. For women of childbearing potential, the result of serum or urine pregnancy test within 7 days prior to the first administration of the study drug shall be negative. If the urine pregnancy test result is positive or cannot be confirmed as negative, a serum pregnancy test shall be required for confirmation.
9. The patient voluntarily participates in the study, signs the informed consent form, and is able to comply with the study schedule for follow-up visits, treatment plans, laboratory tests, and other research procedures.

Exclusion Criteria:

1. A history of malignant tumor is known.
2. Residual toxic reactions caused by prior anti-tumor therapy (including immunotherapy, targeted therapy, chemotherapy, radiotherapy, etc.) (excluding alopecia, fatigue and grade 2 hypothyroidism), or clinically significant laboratory test abnormalities > grade 1 (CTCAE v5.0)
3. Known to have active central nervous system metastases and/or carcinomatous meningitis. Patients with treated brain metastases may participate in the study, provided that their disease is stable.
4. A history of severe hypersensitivity reactions to taxanes or other monoclonal antibodies.
5. Has any contraindication to the study drugs of this project (docetaxel, nimotuzumab, and camrelizumab)
6. Uncontrolled pleural, peritoneal, pelvic or pericardial effusion requiring drainage at least once a month.
7. Uncontrolled or poorly controlled heart diseases, including a history of congestive heart failure (CHF) ≥ Grade 2 (per CTCAE v5.0 or NYHA classification), myocardial infarction, unstable angina pectoris, ventricular tachycardia or torsades de pointes within 6 months prior to enrollment, or cardiac arrhythmias requiring treatment, such as complete left bundle branch block or third-degree atrioventricular block.
8. Pulmonary embolism or deep vein thrombosis occurring within 3 months prior to the first administration of the study drug (excluding catheter-related thrombosis from implanted ports or PICC lines)
9. A history of or current interstitial pneumonia, severe chronic obstructive pulmonary disease complicated with respiratory failure, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
10. Any severe or uncontrolled systemic diseases, including uncontrolled or poorly controlled hypertension (e.g., systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg), diabetes mellitus (glycated hemoglobin (HbA1c) > 8%), etc.
11. Patients with active bleeding, a history of coagulation disorders, or those receiving coumarin anticoagulant therapy.
12. Known to have active hepatitis B or hepatitis C.
13. Complicated with severe, uncontrolled infections, or known human immunodeficiency virus (HIV) infection (positive for HIV antibodies), or diagnosed with acquired immunodeficiency syndrome (AIDS); or with uncontrolled autoimmune diseases; or with a history of allogeneic tissue/organ transplantation, stem cell or bone marrow transplantation, or previous solid organ transplantation.
14. Active bacterial, viral, fungal, rickettsial, or parasitic infections receiving systemic anti-infective therapy (unless treated and resolved prior to the administration of the study drug)
15. Live virus vaccines administered within 30 days prior to the first dose of the study drug. The use of inactivated seasonal influenza vaccines or approved COVID-19 vaccines is permitted, provided that the interval between vaccination and the first dose of the study drug is more than 1 week.
16. Receiving immunology-based therapy for any reason
17. Pregnant or lactating female patients.
18. Any other diseases, clinically significant laboratory parameter abnormalities, severe medical or psychiatric illnesses/conditions, or substance abuse including alcoholism that, in the investigator's judgment, may compromise patient safety, study integrity, affect patient participation in the study, or interfere with the study objectives and outcome analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Imaging assessment after completion of the first 4-6 cycles of therapy (i.e.,at12-18weeks)

SECONDARY OUTCOMES:
For CPS ≥20 and the Overall Population: Median Overall Survival (mOS) | At least up to 24 months.
  mOS is defined as the time from from Day 1 of treatment initiation until death from any cause. mOS corresponds to the time point at which the Kaplan-Meier curve of overall survival probability reaches 50%, estimated using non-parametric interpolation. This endpoint will be analyzed in months.
For CPS ≥20 and the Overall Population: Median Progression-Free Survival (mPFS) | At least up to 24 months.
  mPFS is defined as the time from Day 1 of treatment initiation until the first occurrence of disease progression (per RECIST v1.1), or death from any cause. mPFS corresponds to the time point at which the Kaplan-Meier curve of progression-free survival probability reaches 50%, estimated using non-parametric interpolation. This endpoint will be analyzed in months.
PFS rates at 6 and 12 months | PFS rates at 6 months and 12 months will be recorded separately.
  PFS is defined as the time from the day of first study drug administration to tumor progression (in any aspect) or death (from any cause). PFS rates at 6 months and 12 months will be recorded separately.
Duration of Response (DoR) | At least up to 24 months.
  Defined as the time interval from the first documented complete response (CR) or partial response (PR) per RECIST v1.1 criteria until disease progression or death (whichever occurs earlier). Units are days or months (e.g.,days or months).
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | At least up to 24 months.
  Throughout this study and during the follow-up period, the severity of adverse events will be graded according to NCI-CTCAE v5.0. Safety evaluation metrics include:
  Incidence, severity, and relationship to the study drug of:
  All Adverse Events (AE) Treatment-Emergent Adverse Events (TEAE) Serious Adverse Events (SAE) Immune-Related Adverse Events (irAE).
Quality of Life (QoL) | Baseline, at the end of cycles 2 or 3 (each cycle is 21 days), at the end of cycles 4 or 6 (each cycle is 21 days), and within one week after the final treatment.
  The QoL was assessed at baseline and during follow-up using the EORTC Quality of Life Questionnaire Core 30 (QLQ-C30), Version 3.0, which represent functions, symptoms, or health conditions. The EORTC QLQ-C30: a quality of life instrument for use in international clinical trials in oncology. A total of 30 items are included. Each item is graded from 1 to 4, except for items 29 and 30, indicating not at all, a little, quite a bit, and very much, with higher scores indicating poorer quality of life.
Psychological Scales Assessment as assessed by the Depression, Anxiety, and Stress Scale (DASS-21) | Baseline, at the end of cycles 2 or 3 (each cycle is 21 days), at the end of cycles 4 or 6 (each cycle is 21 days), and within one week after the final treatment.
  Each of the three DASS-21 scales contains 7 items, divided into subscales with similar content. The depression scale assesses dysphoria, hopelessness, devaluationoflife, self-deprecation, lack of interest/involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale is sensitive to levels of chronic non specific arousal.
  Recommended cut-off scores for conventional severity labels（normal,moderate,severe) are as follows: NB Scores on the DASS-21 will need to be multiplied by 2 to caculate the final score:
  Depresslon: normal:0-9, mild:10-13, moderate:14-20, severe: 21-27, extremely severe: 28+.
  Anxlety: normal:0-7, mild: 8-9, moderate:10-14, severe: 15-19, extremely severe: 20+.
  Stress: normal: 0-14, mild: 15-18, moderate:19-25, severe: 26-33, extremely severe:34+.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No